CLINICAL TRIAL: NCT06455982
Title: Effect of a Reduced Carbohydrates Menu Combined With a Ketogenic Supplement on Energy Metabolism in a Senior Residence: the SAGE-2 Study
Brief Title: Reduced Carbohydrates + Ketogenic Supplement on Energy Metabolism
Acronym: SAGE-2
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Université de Sherbrooke (Other)
Collaborators: Nestlé Health Science (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 2025-5533
Record Dates: First submitted 2024-06-06; First posted 2024-06-13 (Actual); Last update posted 2024-06-13 (Actual); Status verified 2024-06

CONDITIONS: Healthy Aging
Keywords: Nutritional intervention; Glucose monitoring; Reduced carb diet; Energy metabolism; Ketones
MeSH Terms: conditions — Ketosis

STUDY DESIGN:
Intervention Model Description: Participants will be compared to themselve (i.e. pre-intervention and post-intervention) The intervention will be 2 months of reduced carbohydrate menu combined with a ketogenic supplement (MCT)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Delta of before/after the intervention (Experimental): 2 months of reduced carbohydrate menu combined with a ketogenic MCT supplement
  Interventions: Dietary Supplement: reduced carbohydrate menu combined with ketogenic supplement

INTERVENTIONS:
Dietary Supplement: reduced carbohydrate menu combined with ketogenic supplement — Participants will eat a reduced carb menu for 2 months and they will take 15g of MCT in the morning and the evening for a total of 30g per day.
  Other Names: RCHO+MCT

SUMMARY:
The present study will evaluate the effects on glucose, ketones and other blood biomarkers, cognition, quality of life, physical activity and well-being of a reduced carbohydrate diet paired with a ketogenic product for 2 months in a population living in a senior residence. This study follows the KetoHome (fall 2022) and SAGE (fall 2023) projects which assessed the feasibility, acceptability and effectiveness of a reduced carbohydrate intervention alone.

ELIGIBILITY:
Inclusion Criteria:

* Older men or women in a senior residence;
* Understand, read and write French;
* Have sufficient visual and hearing acuity to pass cognitive tests;
* Available during the intervention period

Exclusion Criteria:

* Body mass index < 20;
* T1 diabetic;
* T2 insulin-dependent diabetic;
* MMSE < 20;
* Weight loss >10% in the last 6 months involuntary or voluntary;
* Known and uncontrolled hypoglycemia;
* Moderate to severe digestive illnesses that can be aggravated by dietary changes;
* Severe dysphagia;
* Supplementation with MCT oil, ketone salts, ketone esters, adherence to the ketogenic diet, reduced carbohydrate diet, intermittent fasting or other diet or supplements that can significantly increase ketones in the last month;
* Participation in other interventional research projects on nutrition or aimed at metabolic change simultaneously.
* Medical condition that could prevent the participant from completing the study in the opinion of the doctor

Min Age: 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2024-09-05 (Estimated); Primary Completion 2024-12-15 (Estimated); Study Completion 2025-12-15 (Estimated)

PRIMARY OUTCOMES:
Plasma glucose concentration | 2 months
  To evaluate the possible improvement in mean glucose concentration following a reduction in carbohydrates combined with an MCT supplement in people living in a senoir residence for 2 months.
Plasma ketones concentration | 2 months
  To evaluate the possible improvement in mean ketones concentration following a reduction in carbohydrates combined with an MCT supplement in people living in a senoir residence for 2 months.
Plasma insulin concentration | 2 months
  To evaluate the possible improvement in mean insulin concentration following a reduction in carbohydrates combined with an MCT supplement in people living in a senoir residence for 2 months.

SECONDARY OUTCOMES:
Plasma triglycerides concentration | 2 months
  To evaluate the possible improvement in mean triglycerides concentration following a reduction in carbohydrates combined with an MCT supplement in people living in a senoir residence for 2 months.
Plasma cholesterol concentration | 2 months
  To evaluate the possible improvement in mean cholesterol concentration following a reduction in carbohydrates combined with an MCT supplement in people living in a senoir residence for 2 months.

CONTACTS AND LOCATIONS:
Locations (1):
- Centre de recherche sur le vieillissement, Sherbrooke, Quebec, Canada